CLINICAL TRIAL: NCT00306345
Title: Outreach: A Programme for Early Recognition, Quick Response and Timely Treatment of Critically Ill Patients in a University Hospital
Brief Title: Outreach: A Programme for Timely Treatment of Critically Ill Patients in a University Hospital
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Radboud University Medical Center (Other)
Other Study IDs: 001; CMO 301
Record Dates: First submitted 2006-03-22; First posted 2006-03-23 (Estimated); Last update posted 2007-07-12 (Estimated); Status verified 2007-02

CONDITIONS: Patient Centered Care; Postoperative Care; Critical Illness
Keywords: Outreach; Major general surgery; Intensive care; Serious adverse events
MeSH Terms: conditions — Critical Illness | interventions — Community-Institutional Relations

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective

INTERVENTIONS:
Behavioral: Outreach

SUMMARY:
The identification of patients with potential early organ failure is the key in preventing admission or readmission to a critical care facility. The primary goal of the Outreach Project is to ensure that all patients with threatening organ failure receive appropriate and timely treatment in a suitable area; avoid admission to the intensive care unit (ICU); and share ICU skills by a partnership in education. The objectives of the study are to determine whether the introduction of an intensive care unit based medical emergency team, responding to hospital-wide preset criteria of physiologic instability, will decrease the number of predefined serious adverse events (SAEs) and to investigate the effects on quality of life and costs in a general surgery population.

Study Hypothesis: The Outreach intervention will decrease the number of predefined serious adverse events; increase quality of life; and decrease costs.

DETAILED DESCRIPTION:
DESIGN: A multi centre longitudinal intervention trial with a before and after design in a university hospital.

The INTERVENTION consists of three parts:

1. The introduction of a hospital-wide intensive care unit based medical emergency team to evaluate and treat patients deemed at risk for developing an adverse outcome.
2. Education and training of ward staff in the recognition and basic management of patients developing a critical illness.
3. The development of an intensive care (nurse and physician staffed) consultancy service for general wards.

STUDY POPULATION: The population for this study consists of patients undergoing major general surgery with an admission stay of more than 48 hours. It includes patients undergoing central or peripheral vascular surgery, major oncological surgery, lung surgery, major abdominal surgery and trauma surgery.

MEASUREMENTS AND OUTCOMES: In total, 1500 patients will be included. (750 Patients in the control period and 750 patients in the intervention period). Measurements include the incidence of Serious Adverse Events, HRQoL (Quality of life EQ-5D), costs of care and ICU logistics.

TIME-SCHEDULE: Data collection starts January 1, 2006 and stops no later than three months after the inclusion of 1500 patients or April 1, 2008. The final report of the study will be in December 2008.

ELIGIBILITY:
Inclusion Criteria:

* Major general surgery.
* Admitted to the hospital 48 hours after surgical intervention

Exclusion Criteria:

* Not able to communicate in the Dutch language.
* Younger than 18 years old.
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1500 (Estimated)
Dates: Start 2006-01; Study Completion 2008-12

CONTACTS AND LOCATIONS:
Overall Officials: Hans van der Hoeven, Professor, Principal Investigator — UMCN
Locations (1):
- Radboud Universiteit Nijmegen Medical Center, Nijmegen, Gelderland, Netherlands

REFERENCES:
- [Background] Bellomo R, Goldsmith D, Uchino S, Buckmaster J, Hart G, Opdam H, Silvester W, Doolan L, Gutteridge G. Prospective controlled trial of effect of medical emergency team on postoperative morbidity and mortality rates. Crit Care Med. 2004 Apr;32(4):916-21. doi: 10.1097/01.ccm.0000119428.02968.9e. PMID 15071378
- [Background] Hillman K, Chen J, Cretikos M, Bellomo R, Brown D, Doig G, Finfer S, Flabouris A; MERIT study investigators. Introduction of the medical emergency team (MET) system: a cluster-randomised controlled trial. Lancet. 2005 Jun 18-24;365(9477):2091-7. doi: 10.1016/S0140-6736(05)66733-5. PMID 15964445
- [Background] DeVita MA, Bellomo R, Hillman K. Introduction to the rapid response systems series. Jt Comm J Qual Patient Saf. 2006 Jul;32(7):359-60. doi: 10.1016/s1553-7250(06)32046-6. No abstract available. PMID 16884121
- [Background] Devita MA, Bellomo R, Hillman K, Kellum J, Rotondi A, Teres D, Auerbach A, Chen WJ, Duncan K, Kenward G, Bell M, Buist M, Chen J, Bion J, Kirby A, Lighthall G, Ovreveit J, Braithwaite RS, Gosbee J, Milbrandt E, Peberdy M, Savitz L, Young L, Harvey M, Galhotra S. Findings of the first consensus conference on medical emergency teams. Crit Care Med. 2006 Sep;34(9):2463-78. doi: 10.1097/01.CCM.0000235743.38172.6E. PMID 16878033